CLINICAL TRIAL: NCT05648383
Title: An Intersectoral Innovative Solution Involving DIGItal Tools, Empowering Families and Integrating Community CARE Services for the Prevention and Management of Type 2 Diabetes and Hypertension
Brief Title: Promote Health With Digital Tools Among Adults With Type 2 Diabetes/Prediabetes and/or Hypertension
Acronym: DigiCare4You
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harokopio University (Other)
Collaborators: Medical University of Varna (Other); Centre for Research and Technology Hellas (Other); University of Medicine, Tirana (Other); La Trobe University (Other); National and Kapodistrian University of Athens (Other); NYU Langone Health (Other); University Ghent (Other); Universidad de Zaragoza (Other); PRIVANOVA SAS (Unknown); Monash University (Other); METEDA SRL (Unknown); Baker Heart and Diabetes Institute (Other); Sant'Anna School of Advanced Studies (Unknown); International Diabetes Federation (Other); STICHTING INTERNATIONAL FOUNDATION FORINTEGRATED CARE (Unknown); EUROPEAN UNION'S HORIZON 2020 RESEARCH AND INNOVATION PROGRAMME (Project Number: 945246) (Unknown)
Responsible Party: Principal Investigator, Yannis Manios, Professor, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 945246
Record Dates: First submitted 2022-11-28; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Type 2 Diabetes; PreDiabetes; Hypertension
Keywords: community; primary healthcare; families; m-health application; diabetes; hypertension; screening; lifestyle intervention; self-management; people-centred care; scaling-up
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Hypertension; Diabetes Mellitus | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pre-diabetes group, mHealth intervention (Experimental): Participants will receive mHealth intervention (mobile apps) and counseling sessions along with standard care
  Interventions: Behavioral: mHealth intervention
- Diabetes group, mHealth intervention (Experimental): Participants will receive mHealth intervention (mobile apps) and counseling sessions along with standard care
  Interventions: Behavioral: mHealth intervention
- Prediabetes group, control (Active Comparator): Participants will receive standard care, including lifestyle recommendations
  Interventions: Behavioral: Standard care
- Diabetes group, control (Active Comparator): Participants will receive standard care, including lifestyle recommendations
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: mHealth intervention — Participants will receive mHealth intervention (mobile apps) and counseling sessions along with standard care
  Arms: Diabetes group, mHealth intervention; Pre-diabetes group, mHealth intervention
Behavioral: Standard care — Participants will receive standard care, including lifestyle recommendations.
  Arms: Diabetes group, control; Prediabetes group, control

SUMMARY:
The DigiCare4You project will use digital tools for early screening, prevention and management of type 2 diabetes (T2D) and hypertension (HTN). An implementation study will be conducted, targeting more than 10,000 families in two Middle Income Countries (Albania and Bulgaria) and two High Income Countries (Greece and Spain), considering vulnerable groups. Schools will be used as an entry point to the community. Building on an existing procedure for children's periodic growth assessment, conducted by school nurses or in collaboration with local community health centers, parents/ caregivers will be screened via a non-invasive self-reported digital screening tool. Those identified at high risk for T2D will be referred for glycaemia testing (fasting plasma glucose and glycated hemoglobin, HbA1c), as well as blood pressure (BP) measurements, at local community health centers. Parents/ caregivers confirmed to have pre-diabetes or diabetes (and possibly high BP) will be invited to join a mHealth self-management intervention coordinated by the community healthcare workforce. The goal of this intervention is to involve high-risk adults in the treatment process and decision-making on personalized behavioral goals (e.g. diet, physical activity, smoking, alcohol, medication compliance) that meet their needs, and ultimately improve the health status of parents/caregivers, as well as the lifestyle of the entire family.

DETAILED DESCRIPTION:
The rising burden of diabetes poses important public health challenges to health systems nowadays. The age-standardized rates of diabetes prevalence have stabilized in many European countries in recent years, especially in the Nordic countries, but they have gone up in Southern, Eastern and Central EU countries. However, in the vast majority of countries, national diabetes plans are poorly (or not) implemented and underfunded and although T2D is preventable, its prevalence is expected to reach 66 million by 2030, and 68 million by 2045. According to the World Health Organization (WHO)'s "Framework on integrated people-centred health services", integrated people-centred health services put people and communities, not diseases, at the centre of health systems, and empower people to take charge of their own health rather than being passive recipients of services. People-centred care is one of the main goals of health systems, and it is oriented towards the needs of people and their involvement in the treatment process and decision-making. This is expected to result in better care as experienced by people, less inequality, health promotion, better disease prevention, and treatments targeted to people's needs. Health system transition to people-centred care requires empowering citizens and integration of services. The growing digital transformation of health and care offers great opportunity to achieve this transition. Innovative solutions involving digital tools have the potential to improve people-centred care through self-management, goal orientation and shared decision-making. The DigiCare4You project is in line with the WHO's conceptual framework, and is oriented to health promotion and disease prevention through empowering families and integrating care services in local communities to deliver people-centred care for the prevention and management of T2D and HTN. Ultimately, the DigiCare4You project aims to involve high-risk adults in the treatment process and decision-making on personalized behavioral goals (e.g. diet, physical activity, smoking, alcohol, medication compliance) that meet their needs.

The DigiCare4You project proposes a people-centered health service model to prevent and manage T2D and HTN by using the existing resources and adding digital tools for empowering both the existing healthcare workforce and the healthcare recipients. The proposed model aims to integrate two fragmented primary care services, i.e., (a) the children's growth and development monitoring and (b) the early screening and prevention of T2D and HTN. The first one is implemented across all countries in Europe from birth through late adolescence, it includes a physical examination (eye, oral and hearing), anthropometric measurements (weight and height), vaccination evaluation and a brief family medical history, and it is usually linked with the school (primary and secondary education). The latter primary care service related to the screening and prevention of T2D and HTN among the adult population in Europe is poorly or not implemented at all despite the fact that the majority of European countries have made progress towards developing a national plan addressing diabetes specifically or in an overarching plan for non-communicable diseases (NCDs). Integrating the existing children's' growth assessment procedure with the adult screening procedure for NCDs, can help identify and treat parents (and eventually families) at risk for T2D.

Specifically, the proposed model, called DigiCare4You solution, consists of two core components: a) a two-stage systematic screening procedure, and (b) a mHealth, community-based intervention. The two-stage screening procedure will be implemented using schools as the entry point to the community in order to reach as many parents with children at primary or secondary education as possible, and assess their risk for T2D and/or HTN. First, high risk parents will be identified through a digitalized non-invasive screening procedure (1st stage screening), using a self-reported questionnaire, the Finnish Diabetes Risk Score (FINDRISC). Those parents with a FINDRISC ≥10 will be referred to glycaemia testing (i.e., fasting plasma glucose [FPG], and glycated hemoglobin [HbA1c]) according to the national guidelines in each country) and blood pressure evaluation (2nd stage screening). Parents confirmed to have pre-diabetes or diabetes will be invited to join the self-management intervention including access to the DigiCare4You mHealth applications. The DigiCare4You mHealth applications will assist users make personalised decisions with respect to behavioral changes (e.g., diet tracking and meal planning, physical activity, sleep quantity), medication use (if applicable), scheduling/reminding re-examination visits and prospectively monitoring their health outcomes. Last but not least, these applications will enable direct communication between the users and their healthcare providers through feedback messages and reports, including lab results.

DigiCare4You acknowledges the differences in health and care systems across Europe and considering the vulnerable and underserved groups, will be adapted and implemented in two Middle-income countries (MICs), Albania and Bulgaria, and two High-income countries (HICs), Greece and Spain, all with high prevalence of T2D and HTN and weak primary healthcare systems. Furthermore, in all countries, both municipalities of medium-high and low socioeconomic status (SES) areas (with low literacy levels, high rates of unemployment and large proportions of immigrants) will also be included. Overall, the DigiCare4You solution will ensure that even the most underserved parts of the community will be reached and any potential barrier towards achieving equal access for all will be tackled. This approach will allow the evaluation of the success and validity of the solution among MICs and HICs, and among the underserved and marginalized populations within countries. Therefore, if the DigiCare4You solution will be proven to be equally effective among high and low-SES groups, this will ensure that the uptake of the solution at large scale will promote equity in health and easy access to primary healthcare services for the overall population. A hybrid II implementation study will be designed to implement and evaluate the DigiCare4You solution, comparing the mHealth intervention (intervention arm) with the existing standard care (control arm). In all four countries, a 1:1 cluster-randomized design will be followed, randomly allocating municipalities (therefore the schools, the local community health centers and the families within each municipality) to either the intervention or the control arm. DigiCare4You intervention will have a two-year duration and all measurements for the impact and outcome evaluation will take place at baseline and at 12- and 24-months follow-ups, while the process evaluation at participant, school and community level will be ongoing throughout the implementation period.

ELIGIBILITY:
Inclusion Criteria:

* People who have their permanent residence within the prefecture/region of the relevant facility participating in the clinical study.
* People having children at primary and/ or secondary education.
* People who are physically and mentally able to provide their informed consent to participate.
* People with a FINDRISC ≥10
* People with a fasting plasma glucose (FPG) ≥ 100 mg/dL and /or glycated hemoglobin (HbA1c) ≥ 5.7%

Exclusion Criteria:

* People suffering from a health condition where adherence to the intervention will be contraindicated or improbable.
* People unable to express a free and informed consent for medical and/or psychological conditions, mental incapacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 992 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in fasting plasma glucose [FPG] at 12 months (1st follow-up) | Baseline and 12 months (1st follow-up)
  Fasting plasma glucose [FPG] is measured in participants with T2D and in participants with prediabetes at 12 months (1st follow-up) from baseline.
Change from Baseline in fasting plasma glucose [FPG] at 24 months (2nd follow-up) | Baseline and 24 months (2nd follow-up)
  Fasting plasma glucose [FPG] is measured in participants with T2D and in participants with prediabetes at 24 months (2nd follow-up) from baseline.
Change from Baseline in glycated hemoglobin [HbA1c] at 12 months (1st follow-up) | Baseline and 12 months (1st follow-up)
  Glycated hemoglobin [HbA1c] is measured in participants with T2D and in participants with prediabetes at 12 months (1st follow-up) from baseline.
Change from Baseline in glycated hemoglobin [HbA1c] at 24 months (2nd follow-up) | Baseline and 24 months (2nd follow-up)
  Glycated hemoglobin [HbA1c] is measured in participants with T2D and in participants with prediabetes at 24 months (2nd follow-up) from baseline.

SECONDARY OUTCOMES:
Change from Baseline in blood pressure [BP] at 12 months (1st follow-up) | Baseline and 12 months (1st follow-up)
  Blood pressure [BP] is measured in participants with T2D and in participants with prediabetes at 12 months (1st follow-up) from baseline.
Change from Baseline in blood pressure [BP] at 24 months (2nd follow-up) | Baseline and 24 months (2nd follow-up)
  Blood pressure [BP] is measured in participants with T2D and in participants with prediabetes at 24 months (2nd follow-up) from baseline.
Change from Baseline in body weight [BW] at 12 months (1st follow-up) | Baseline and 12 months (1st follow-up)
  Body weight [BW] is measured in participants with T2D and in participants with prediabetes at 12 months (1st follow-up) from baseline.
Change from Baseline in body weight [BW] at 24 months (2nd follow-up) | Baseline and 24 months (2nd follow-up)
  Body weight [BW] is measured in participants with T2D and in participants with prediabetes at 24 months (2nd follow-up) from baseline.
Change from Baseline in waist circumference [WC] at 12 months (1st follow-up) | Baseline and 12 months (1st follow-up)
  Waist circumference [WC] is measured in participants with T2D and in participants with prediabetes at 12 months (1st follow-up) from baseline.
Change from Baseline in waist circumference [WC] at 24 months (2nd follow-up) | Baseline and 24 months (2nd follow-up)
  Waist circumference [WC] is measured in participants with T2D and in participants with prediabetes at 24 months (2nd follow-up) from baseline.

OTHER OUTCOMES:
Change form Baseline in the BMI z-score of children at 12 months (1st follow-up) | Baseline and 12 months (1st follow-up)
  Although children will not directly receive any intervention, their BMI z-score will be calculated at 12 months (1st follow-up) of the intervention in parents with T2D and in parents with prediabetes. Change = (Month 12 score - Baseline score)
Change form Baseline in the BMI z-score of children at 24 months (2nd follow-up) | Baseline and 24 months (2nd follow-up)
  Although children will not directly receive any intervention, their BMI z-score will be calculated at 24 months (2nd follow-up) of the intervention in parents with T2D and in parents with prediabetes. Change = (Month 24 score - Baseline score)

CONTACTS AND LOCATIONS:
Overall Officials: Yannis Manios, Professor, Principal Investigator — Harokopio University
Locations (4):
- Universiteti i Mjekësisë, Tirana, Rruga E Dibrës, Albania
- Medical University of Varna, Varna, Bulgaria
- Harokopio University, Athens, Attica, Greece
- Universidad de Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared with the project partners and third parties.Although a preliminary version of the Data Management Plan has been developed, there are still a few points to be finalized, including the time frame with respect to data availability, the access criteria regarding how requests for information will be reviewed, and if a web address will be used to share IPD.
Time Frame: This has not been decided yet.
Access Criteria: For the duration of the project, data will be stored in a Secure Cloud-Based Repository, managed by the Project Coordinator who will authorize access to project partners' staff; when partners or partners' staff leave the project, the access to the repository will be disabled. Third parties will be granted access to the data for research purposes, including validation of the results presented in scientific publications.

REFERENCES:
- [Result] Manios Y, Mavrogianni C, Lambrinou CP, Cardon G, Lindstrom J, Iotova V, Tankova T, Civeira F, Kivela J, Jancso Z, Shadid S, Tsochev K, Mateo-Gallego R, Rado S, Dafoulas G, Makrilakis K, Androutsos O; Feel4Diabetes-study group. Two-stage, school and community-based population screening successfully identifies individuals and families at high-risk for type 2 diabetes: the Feel4Diabetes-study. BMC Endocr Disord. 2020 Mar 12;20(Suppl 1):12. doi: 10.1186/s12902-019-0478-9. PMID 32164646
- [Result] Manios Y, Androutsos O, Lambrinou CP, Cardon G, Lindstrom J, Annemans L, Mateo-Gallego R, de Sabata MS, Iotova V, Kivela J, Martinez R, Moreno LA, Rurik I, Schwarz P, Tankova T, Liatis S, Makrilakis K. A school- and community-based intervention to promote healthy lifestyle and prevent type 2 diabetes in vulnerable families across Europe: design and implementation of the Feel4Diabetes-study. Public Health Nutr. 2018 Dec;21(17):3281-3290. doi: 10.1017/S1368980018002136. Epub 2018 Sep 12. PMID 30207513
- [Result] Lindstrom J, Tuomilehto J. The diabetes risk score: a practical tool to predict type 2 diabetes risk. Diabetes Care. 2003 Mar;26(3):725-31. doi: 10.2337/diacare.26.3.725. PMID 12610029
- [Result] Mavrogianni C, Lambrinou CP, Androutsos O, Lindstrom J, Kivela J, Cardon G, Huys N, Tsochev K, Iotova V, Chakarova N, Rurik I, Moreno LA, Liatis S, Makrilakis K, Manios Y; Feel4Diabetes-study group. Evaluation of the Finnish Diabetes Risk Score as a screening tool for undiagnosed type 2 diabetes and dysglycaemia among early middle-aged adults in a large-scale European cohort. The Feel4Diabetes-study. Diabetes Res Clin Pract. 2019 Apr;150:99-110. doi: 10.1016/j.diabres.2019.02.017. Epub 2019 Feb 20. PMID 30796939
- [Result] Oldenburg B, Taylor CB, O'Neil A, Cocker F, Cameron LD. Using new technologies to improve the prevention and management of chronic conditions in populations. Annu Rev Public Health. 2015 Mar 18;36:483-505. doi: 10.1146/annurev-publhealth-031914-122848. Epub 2015 Jan 12. PMID 25581147
- [Result] O'Neil A, Cocker F, Rarau P, Baptista S, Cassimatis M, Barr Taylor C, Lau AYS, Kanuri N, Oldenburg B. Using digital interventions to improve the cardiometabolic health of populations: a meta-review of reporting quality. J Am Med Inform Assoc. 2017 Jul 1;24(4):867-879. doi: 10.1093/jamia/ocw166. PMID 28339628
- See also: DigiCare4You link website — https://digicare4you.eu/